CLINICAL TRIAL: NCT06611202
Title: Enhancing Mobility and Mental Health in Dementia Patients: A Multidisciplinary Six-Minute Walking Group Pilot Study
Brief Title: Enhancing Mobility and Mental Health in Dementia Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxleas NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Tolulope Adeniji PhD PT, Dr, Oxleas NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS Project ID: 349221
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Dementia
Keywords: older adult; physical activity; cognitive impairment; mental health
MeSH Terms: conditions — Dementia; Motor Activity; Cognitive Dysfunction; Psychological Well-Being | interventions — Exercise; Walking; Clonazepam

STUDY DESIGN:
Intervention Model Description: Single-group pretest-post-test design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- six minute walking group (Experimental): Intervention:
  Physiotherapy Component: A six-minute walking group will be conducted twice a week for 8 weeks, targeting improvements in mobility, endurance, and balance. Occupational Therapy Intervention: Occupational therapists will integrate functional tasks (Games and throwing of balls to court, bean bag target game to enhance exercise relevance to daily activities. Psychological Support: A psychologist will provide mental health support during the sessions, utilising techniques like time focus reminiscence therapy to engage patients
  Interventions: Other: Exercise; Drug: Clonazepam

INTERVENTIONS:
Other: Exercise — A multidisciplinary six-minute walking group intervention-spearheaded by physiotherapists, occupational therapists, and psychologists-in enhancing physical activity, mobility, cognitive function, and functional independence among patients with dementia.
  Physiotherapy Component: A six-minute walking group will be conducted twice a week for 8 weeks, targeting improvements in mobility, endurance, and balance. Occupational Therapy Intervention: Occupational therapists will integrate functional tasks (Games and throwing of balls to court, bean bag target game to enhance exercise relevance to daily activities. A psychologist will provide mental health support during the sessions, utilising techniques like time focus reminiscence therapy to engage patients and reduce anxiety.
  Other Names: walking; remniscent therapy; functional activities
Drug: Clonazepam — Medication on our dementia wards are being review during ward round and when needs arise. The medication management in drugs will be fully documented and accounted for in the course of the study.

SUMMARY:
This study aims to evaluate the effect of a multidisciplinary six-minute walking group and activities on patients with dementia's physical activity levels, mobility, anxiety, and cognitive function. The primary objective of this study is to evaluate the effectiveness of a multidisciplinary six-minute walking group intervention-spearheaded by physiotherapists, occupational therapists, and psychologists-in enhancing physical activity, mobility, cognitive function, and functional independence among patients with dementia. A systematic review of existing evidence on the effectiveness of the existing interventions will be conducted to contextualise the findings, providing a robust benchmark for assessing the contribution of each therapeutic component.

Secondary Objectives:

1. Physiotherapy Impact: To determine the specific effects of physiotherapy on mobility, endurance, and balance in dementia patients using validated, objective measures.
2. Occupational Therapy Contribution: To evaluate the role of occupational therapy in improving functional independence and the ability to perform daily activities through targeted, task-oriented activities.
3. Psychological Impact: To assess the psychological benefits of the intervention, including reductions in anxiety and enhancements in mood and overall mental health, as a result of the psychologist-led component.
4. Dietary Support Role: To investigate the influence of integrated dietary support on physical activity levels, nutritional status, and overall health.
5. Feasibility and Scalability: To explore the practicality of integrating this multidisciplinary intervention into routine dementia care and assess its potential for broader application across similar settings.

DETAILED DESCRIPTION:
This study aim to implement and evaluate a multidisciplinary intervention designed to enhance mobility level, cognition and physical activity levels in dementia patients within an inpatient ward. Central to this intervention is a six-minute walking group led collaboratively by physiotherapists, occupational therapists (OT), and psychologists. The program will be augmented by tailored nutritional support from dietitians and ongoing psychiatric/medical team consultation. A vital component of this initiative is a scoping review, which will synthesise existing evidence on similar interventions, providing a robust foundation for the studys design and establishing benchmarks for assessing the effectiveness of each therapeutic element. This project will be piloted within one of our dementia ward, this project has significant potential for broader implementation across other units, directly supporting our mission to enhance the 'Culture of Care' by integrating evidence-based practices into the daily care routines of dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dementia.
* Older adults from the age 65 and above
* Must be able to mobilise independently.
* Must be able to engage with minimal tasks that will be based on the

Exclusion Criteria:

* Must be free from acute comorbidities: Heart failure; hearing loss;
* Free from significant visual impairment
* Must be free from orthostatic hypotension

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Mobility | 8 weeks
  A six-minute walking group will be conducted twice a week for 8 weeks, targeting improvements in mobility, endurance, and balance. The impact of physiotherapy will be evaluated using objective tools such as the Tinetti Balance and Gait Assessment. The Tinetti balance subdomain has 16 items, and the gait component has 12 items, with 28 possible outcomes on the tool. The higher the score the better the balance and gait outcome
Mobility | 8 weeks
  A six-minute walking group will be conducted twice a week for 8 weeks, targeting improvements in mobility, endurance, and balance. The impact of physiotherapy will be evaluated using an objective tool called the Elderly Mobility Scale (EMS), with outcomes ranging from 0 to 20. The higher the score the better the mobility level outcome

SECONDARY OUTCOMES:
Functional tasks | 8 weeks
  Occupational therapists will integrate functional tasks, such as ball games involving throwing balls into a court and a bean bag target game, to enhance the relevance of exercises to daily activities. The effectiveness of occupational therapy will be measured by improvements in functional independence using the Pool Activity Level, PAL, Checklist. The Pool Activity Level (PAL) Checklist scores range from 1 to 10, indicating varying degrees of functional independence and engagement in daily activities. A score of 1 to 2 represents profound limitations requiring maximum assistance, while scores of 3 to 4 indicate severe limitations with significant support needed. Moderate independence is reflected in scores of 5 to 6, and scores of 7 to 8 show mild independence, allowing for participation with minimal assistance. Scores of 9 to 10 represent the highest level of independence, where individuals can plan and carry out activities independently. The higher the score the better
mental health and cognition | 8 weeks
  A psychologist will provide mental health support during the sessions, utilising techniques like time focus reminiscence therapy to engage patients and reduce anxiety. The psychological impact will be assessed using the Neuropsychiatric Inventory Questionnaire (NPI-Q). The Neuropsychiatric Inventory Questionnaire, NPI-Q, assesses a range of neuropsychiatric symptoms, with scoring reflecting the severity and frequency of behaviours. Each item is rated based on how often the behaviour occurs from 0 for not at all to 3 for very frequently and the severity of the impact on daily life from 0 for not severe to 3 for very severe. Total scores can range from 0 to 30, with higher scores indicating more significant neuropsychiatric symptoms and a greater psychological impact on the individual. This scoring system helps psychologists evaluate the effectiveness of interventions and tailor support accordingly.
mental health and cognition | 8 weeks
  Therapy team will measure global cognitive function with short version of the IQCODE. The IQCODE short version is a tool used to assess cognitive decline by evaluating an individual's abilities over the past 5 or 10 years. It consists of 16 items, each rated on a scale from one to five, with lower scores indicating better cognitive function. Total scores range from 16 to 80, with higher scores suggesting greater cognitive impairment. The scoring helps identify changes in cognitive abilities and aids in the diagnosis of dementia and other cognitive disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Holbrook ward, Sidcup, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator plan to share individual participant data (IPD) with other researchers. Data will include de-identified participant data that support the results reported in the study. Access will be granted to qualified researchers who submit a request along with a scientifically sound proposal, subject to approval by the data-sharing committee.
Supporting Information: Study Protocol, SAP, ICF